CLINICAL TRIAL: NCT03669029
Title: Optimization of Golimumab Treatment in Ulcerative Colitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Manises (Other)
Collaborators: General University Hospital of Valencia (Other); Hospital Clínico Universitario de Valencia (Other); Hospital de Sagunto (Other); Hospital Universitario La Fe (Other); Hospital General Universitario de Alicante (Other); Hospital Universitario Doctor Peset (Other); Hospital Arnau de Vilanova (Other); Hospital Provincial de Castellon (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JHV-GOL-2018-01
Record Dates: First submitted 2018-07-04; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Colitis, Ulcerative
Keywords: Golimumab; Inflammatory Bowel Disease; Optimization; Drug levels; Anti-drug antibody levels
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Week 6 Responders (Experimental): In patients with clinical response at week 6, serum golimumab levels and anti-golimumab antibody levels will be correlated with clinical response.
  Interventions: Drug: Golimumab 50 mg in patients <80 kg and Golimumab 100 mg in patients >80 kg
- Week 6 Non Responders (Experimental): In patients without clinical response at week 6, golimumab treatment will be optimized.
  Interventions: Drug: Golimumab treatment optimization.

INTERVENTIONS:
Drug: Golimumab 50 mg in patients <80 kg and Golimumab 100 mg in patients >80 kg — Clinical response at week 6,14, 30 and 54 will be correlated to serum golimumab levels and anti-golimumab antibody levels.
  Arms: Week 6 Responders
Drug: Golimumab treatment optimization. — Golimumab dosing will be optimized in patients without clinical response at week 6.
  Arms: Week 6 Non Responders

SUMMARY:
This is a multicenter, prospective study of dose adjustment of golimumab in patients with ulcerative colitis who will initiate golimumab treatment (naïve to anti-TNF) or after failure (or exposure) to one anti-TNF, which aims to analyze serum golimumab levels and anti- golimumab antibody (ADA) levels during the induction (week 6) and maintenance phases (week 14, 30 and 54) and correlate them with efficacy parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years or older, both sexes and any race) who will be treated with Golimumab according to clinical criteria.

Exclusion Criteria:

* Patients with Crohn's disease or colitis pending classification
* Patients with ileoanal pouch
* Patients with perianal fistulas related to the disease
* Patients with a history of hypersensitivity to golimumab, other murine proteins, or to any of the excipients included in the golimumab datasheet.
* Patients with tuberculosis or other serious infections such as septicemia, abscesses and opportunistic infections.
* Patients with moderate or severe heart failure (NYHA grade III / IV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between serum Golimumab levels and clinical response. | Week 6.
  Serum Golimumab levels will be measured and clinical activity evaluation will be assessed according to the partial Mayo score and biochemical parameters such as C-reactive protein and calprotectin.
Correlation between anti-Golimumab antibody levels and clinical response. | Week 6.
  Anti-golimumab antibody levels will be measure and clinical activity evaluation will be performed according to the partial Mayo score and biochemical parameters such as C-reactive protein and calprotectin.

SECONDARY OUTCOMES:
Treatment optimization outcome. | Week 14
  Analyze the percentage of non-responder patients or patients with partial response at week 6 who achieve response/remission at week 14 after treatment optimization.
Correlation between mucosal healing and serum Golimumab levels. | Week 54
  An endoscopy will be performed at the end of the treatment and serum Golimumab levels will be measured.
Identification of cut-off values of serum golimumab concentration | Week 6
  Identify useful cut-off values of serum golimumab concentration for use in ulcerative colitis practice.
Correlation between mucosal healing and anti-Golimumab antibody levels. | Week 54
  An endoscopy will be performed at the end of the treatment and anti-Golimumab antibody levels will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Hinojosa del Val, MD, Principal Investigator — Hospital de Manises
Locations (1):
- Joaquín Hinojosa del Val, Manises, Valencia, Spain

REFERENCES:
- [Background] Dostalek M, Gardner I, Gurbaxani BM, Rose RH, Chetty M. Pharmacokinetics, pharmacodynamics and physiologically-based pharmacokinetic modelling of monoclonal antibodies. Clin Pharmacokinet. 2013 Feb;52(2):83-124. doi: 10.1007/s40262-012-0027-4. PMID 23299465
- [Background] Vande Casteele N, Ballet V, Van Assche G, Rutgeerts P, Vermeire S, Gils A. Early serial trough and antidrug antibody level measurements predict clinical outcome of infliximab and adalimumab treatment. Gut. 2012 Feb;61(2):321; author reply 322. doi: 10.1136/gut.2010.236869. Epub 2011 Feb 17. No abstract available. PMID 21330576
- [Background] Ordas I, Mould DR, Feagan BG, Sandborn WJ. Anti-TNF monoclonal antibodies in inflammatory bowel disease: pharmacokinetics-based dosing paradigms. Clin Pharmacol Ther. 2012 Apr;91(4):635-46. doi: 10.1038/clpt.2011.328. Epub 2012 Feb 22. PMID 22357456
- [Background] Steenholdt C, Al-khalaf M, Brynskov J, Bendtzen K, Thomsen OO, Ainsworth MA. Clinical implications of variations in anti-infliximab antibody levels in patients with inflammatory bowel disease. Inflamm Bowel Dis. 2012 Dec;18(12):2209-17. doi: 10.1002/ibd.22910. Epub 2012 Feb 16. PMID 22344964
- [Background] Fasanmade AA, Adedokun OJ, Blank M, Zhou H, Davis HM. Pharmacokinetic properties of infliximab in children and adults with Crohn's disease: a retrospective analysis of data from 2 phase III clinical trials. Clin Ther. 2011 Jul;33(7):946-64. doi: 10.1016/j.clinthera.2011.06.002. Epub 2011 Jul 7. PMID 21741088
- [Background] Fasanmade AA, Adedokun OJ, Ford J, Hernandez D, Johanns J, Hu C, Davis HM, Zhou H. Population pharmacokinetic analysis of infliximab in patients with ulcerative colitis. Eur J Clin Pharmacol. 2009 Dec;65(12):1211-28. doi: 10.1007/s00228-009-0718-4. Epub 2009 Sep 16. PMID 19756557
- [Background] Sandborn WJ, Feagan BG, Marano C, Zhang H, Strauss R, Johanns J, Adedokun OJ, Guzzo C, Colombel JF, Reinisch W, Gibson PR, Collins J, Jarnerot G, Hibi T, Rutgeerts P; PURSUIT-SC Study Group. Subcutaneous golimumab induces clinical response and remission in patients with moderate-to-severe ulcerative colitis. Gastroenterology. 2014 Jan;146(1):85-95; quiz e14-5. doi: 10.1053/j.gastro.2013.05.048. Epub 2013 Jun 2. PMID 23735746
- [Background] Sandborn WJ, Feagan BG, Marano C, Zhang H, Strauss R, Johanns J, Adedokun OJ, Guzzo C, Colombel JF, Reinisch W, Gibson PR, Collins J, Jarnerot G, Rutgeerts P; PURSUIT-Maintenance Study Group. Subcutaneous golimumab maintains clinical response in patients with moderate-to-severe ulcerative colitis. Gastroenterology. 2014 Jan;146(1):96-109.e1. doi: 10.1053/j.gastro.2013.06.010. Epub 2013 Jun 14. PMID 23770005
- [Background] Adedokun OJ, Xu Z, Marano CW, Strauss R, Zhang H, Johanns J, Zhou H, Davis HM, Reinisch W, Feagan BG, Rutgeerts P, Sandborn WJ. Pharmacokinetics and Exposure-response Relationship of Golimumab in Patients with Moderately-to-Severely Active Ulcerative Colitis: Results from Phase 2/3 PURSUIT Induction and Maintenance Studies. J Crohns Colitis. 2017 Jan;11(1):35-46. doi: 10.1093/ecco-jcc/jjw133. Epub 2016 Jul 20. PMID 27440869
- [Background] Berends S, Strik A, van Egmond P, Brandse H, Mathôt R,D'Haens G, Löwenberg M. Pharmacokinetics of golimumab in patients with moderate tosevere ulcerative colitis. J Crohn´s Colitis 2016; 10 (suppl 1):s424 AP637
- [Background] Hutas G. Berends S, Strik A, van Egmond P, Brandse H, Mathôt R,D'Haens G, Löwenberg M. Pharmacokinetics of golimumab in patients with moderate tosevere ulcerative colitis. J Crohn´s Colitis 2016; 10 (suppl 1):s424 AP637